CLINICAL TRIAL: NCT00330369
Title: DORADO - A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel Group Study to Evaluate the Efficacy and Safety of Fixed Doses of Darusentan in Subjects With Resistant Systolic Hypertension Receiving Combination Therapy With Three or More Antihypertensive Drugs, Including a Diuretic (Protocol DAR-311)
Brief Title: DORADO - Fixed Doses of Darusentan as Compared to Placebo in Resistant Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAR-311
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — darusentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Darusentan Placebo (Placebo Comparator): Placebo to match darusentan for 2-week placebo run-in period, followed by placebo to match darusentan administered orally once daily for 14 weeks
  Interventions: Drug: Darusentan Placebo
- Darusentan 50 mg (Experimental): Placebo to match darusentan for 2-week placebo run-in period, followed by darusentan 50 mg administered orally once daily for 14 weeks
  Interventions: Drug: Darusentan; Drug: Darusentan Placebo
- Darusentan 100 mg (Experimental): Placebo to match darusentan for 2-week placebo run-in period, followed by darusentan 100 mg administered orally once daily for 14 weeks
  Interventions: Drug: Darusentan; Drug: Darusentan Placebo
- Darusentan 300 mg (Experimental): Placebo to match darusentan for 2-week placebo run-in period, followed by darusentan 300 mg administered orally once daily for 14 weeks
  Interventions: Drug: Darusentan; Drug: Darusentan Placebo

INTERVENTIONS:
Drug: Darusentan — Darusentan administered orally once daily
  Other Names: LU 135252
  Arms: Darusentan 100 mg; Darusentan 300 mg; Darusentan 50 mg
Drug: Darusentan Placebo — Placebo to match darusentan administered orally once daily

SUMMARY:
This is a research study of a new experimental drug called darusentan. Darusentan is not currently approved by the U.S. Food and Drug Administration (FDA) for use in the United States, which means that a doctor cannot prescribe this drug. The purpose of this study is to determine if darusentan is effective in reducing systolic blood pressure in subjects with resistant systolic hypertension, despite treatment with full doses of three or more antihypertensive drugs, including a diuretic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are competent to provide written consent
* Aged 35 to 80 years
* Subjects with diabetes and/or chronic kidney disease must have a mean systolic blood pressure ≥130 mmHg
* All other subjects must have a mean systolic blood pressure ≥140 mmHg
* Receiving and adhering to full doses of appropriate guideline-recommended antihypertensive drugs from three different classes of antihypertensive agents, including a diuretic
* Female subjects of non-childbearing potential (i.e., post-menopausal for at lest 2 years; surgically sterile)

Exclusion Criteria:

* Average sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg
* Serum ALT or AST >2 x the upper limit of the normal range (ULN)
* Subjects who have experienced myocardial infarction, unstable angina pectoris, or a cerebrovascular accident (CVA) within 6 month; or sick sinus syndrome or second or third degree atrioventricular block, atrial fibrillation or recurrent atrial tachyarrhythmia, recurrent ventricular tachycardia, or symptomatic bradycardia
* Implanted pacemakers or implanted cardioverter defibrillator (ICD)
* Symptomatic congestive heart failure requiring treatment
* Hemodynamically significant valvular heart disease
* Type I diabetes mellitus
* Hemodialysis or peritoneal dialysis; or history of renal transplant
* Diagnosis or recurrence of malignancy within the past 3 years
* Sleep apnea, unless a recent sleep study demonstrates arterial oxygen saturation greater than or equal to 90%
* Subjects who perform alternating shift or night work
* Subjects who have participated in a clinical study involving another investigational drug or device within 4 weeks prior to Screening

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in trough sitting systolic and diastolic blood pressure measured by sphygmomanometry | Baseline to Week 14

SECONDARY OUTCOMES:
Change from baseline in mean 24-hour systolic and diastolic ambulatory blood pressure | Baseline to Week 14
Percentage of subjects to reach systolic blood pressure goal | Week 14
Change from baseline in estimated glomerular filtration rate (eGFR) | Baseline to Week 14

CONTACTS AND LOCATIONS:
Locations (115):
- United States (67):
  - UAB Hypertension Program, Birmingham, Alabama
  - Comprehensive Heart Failure Center, Mobile, Alabama
  - Canyon Clinical Research, Tucson, Arizona
  - Chrishard Medical Group, Inglewood, California
  - VA Medical Center - WLA, Los Angeles, California
  - Sacramento Heart and Vascular, Sacramento, California
  - Apex Research Institute, Santa Ana, California
  - Complete Renal Care, Denver, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - MedStar Diabetes Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Deerfield Beach Cardiology Associates, Deerfield Beach, Florida
  - White-Wilson Medical Center, Fort Walton Beach, Florida
  - AMK Research, Gainsville, Florida
  - A.G.A. Clinical Trials, Hialeah, Florida
  - Jacksonville Center for Clinical, Jacksonville, Florida
  - Ricardo A. Bedoya, Cardiology, Jupiter, Florida
  - International Research Association, Miami, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Tampa Bay Nephrology, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Global Research Partners, Calhoun, Georgia
  - Kula Research, Honolulu, Hawaii
  - Chicago Heart & Vein Clinic, Elk Grove Village, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - American Clinical Research LLC, Marrero, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Cardiovascular Consultants of Maine, Scarborough, Maine
  - MODEL Clinical Research, Baltimore, Maryland
  - Maryland Medical Research/Og Medical Center, Oxon Hill, Maryland
  - Clinical Associates, Reisterstown, Maryland
  - Rockville Internal Medicine Group, Rockville, Maryland
  - Professional Clinical Research, Benzonia, Michigan
  - Nephrology and Hypertension / Hurley Medical Center, Flint, Michigan
  - Professional Clinical Research, Interlochen, Michigan
  - Specialty Medical Center, Pahrump, Nevada
  - Bronx VA Medical Center / Mt. Sinai, The Bronx, New York
  - Physicians East, PA, Greenville, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - West Coast Cardiology Associates, Fairview Park, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - Southwest Cardiology Associates, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, Tulsa, Oklahoma
  - Hillsboro Cardiology, PC, Hillsboro, Oregon
  - Northeast Clinical Research Centers, Inc., Allentown, Pennsylvania
  - Heritage Cardiology Associates, Camp Hill, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - RI Hospital, Providence, Rhode Island
  - Neem Research Group, Inc., Columbia, South Carolina
  - Internal Medicine & Industrial Medicine, DeSoto, Texas
  - T&R Clinical, P.A., Fort Worth, Texas
  - Pri-Med Care, Lewisville, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Diabetes Center of the Southwest, Midland, Texas
  - The Bracane Company, Plano, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Burke Internal Medicine, Inc., Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Peninsula Inernal Medicine, Gig Harbor, Washington
  - Liberty Research Center, Tacoma, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
- Argentina (10):
  - CIMEL, Buenos Aires
  - DIM (Clinica Privada), Buenos Aires
  - Fundapres, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital Jose Maria Ramos Meijia, Buenos Aires
  - Hospital Municipal bernardo Houssay, Buenos Aires
  - Medeos, Buenos Aires
  - Sanatorio Municipal Dr. Julio Mendez, Buenos Aires
  - Clinica Chutro SRL, Córdoba
  - Hospital San Roque, Córdoba
- Brazil (10):
  - Hospital Governador Israel Pinheiro, Belo Horizonte
  - Hospital Socor, Belo Horizonte
  - Centro Medico de Campinas, Campinas
  - Hospital de Clinicas da Universidade Federal do Parana, Curitiba
  - Hospital das Clinicas, Goiânia
  - Clinica de Exames, Maceió
  - Instituto de Molestias, São José do Rio Preto
  - Centro Integrado Hospital do Rim e Hipertensao, São Paulo
  - Centro integrado hospital, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP, São Paulo
- Canada (2):
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Clinical Research Solutions, Kitchener, Ontario
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Hvidovre Hospital, Hvidovre
- France (5):
  - CIC Hopital Jeanne D'Arc, Dommartin-lès-Toul
  - CHU de Grenoble, Grenoble
  - CHU la Timone Service de cardiologie, Marseille
  - CHU Victor Provo, Roubaix
  - Hôpital Civil, Service HTA maladies vasculaires, Strasbourg
- Germany (5):
  - Kerckhoff-Klinik Forschungs GmbH, Bad Nauheim
  - Charité Campus Buch, Berlin
  - St Josefs-Hospital, Cloppenburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Lübeck
- Azienda Ospedaliera University of Padua Policlinico, Padua, Italy
- Spain (8):
  - Hospital Universitario de Santiago, A Coruña
  - Fundacio Puigvert, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clínico San Cecilio, Granada
  - Hospital Clínico de San Carlos, Madrid
  - Hospital Universitario 12 de Octobre, Madrid
  - Hospital Carlos Haya, Málaga
- Cardiovascular Research, Karolinska Institue, Stockholm, Sweden
- United Kingdom (4):
  - Stonehill Medical Centre, Bolton
  - Townhead Surgery, Scotland
  - Avenue Surgery, Wiltshire
  - Hathaway Medical Centre, Wiltshire

REFERENCES:
- [Derived] Weber MA, Black H, Bakris G, Krum H, Linas S, Weiss R, Linseman JV, Wiens BL, Warren MS, Lindholm LH. A selective endothelin-receptor antagonist to reduce blood pressure in patients with treatment-resistant hypertension: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Oct 24;374(9699):1423-31. doi: 10.1016/S0140-6736(09)61500-2. Epub 2009 Sep 11. PMID 19748665
- See also: Related Info — http://www.gilead.com